CLINICAL TRIAL: NCT00613249
Title: A Double-Blind, Randomized, Placebo-Controlled Phase I Study to Compare the Pharmacokinetics of Intravaginal Dapivirine Gel 4750, 0.05%, 2.5g and Dapivirine Gel 4789, 0.05%, 2.5g Formulations and to Assess the Safety as Compared to the Intravaginal HEC-Based Universal Placebo Gel, 2.5g in Healthy HIV-Negative Women.
Brief Title: A Phase I Pharmacokinetics and Safety Study of Two Dapivirine Intravaginal Gels
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Dr. Annalene Nel, International Partnership for Microbicides
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IPM 012
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2009-03-27 (Estimated); Status verified 2009-03

CONDITIONS: HIV Infections
Keywords: HIV-1 Infection; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Drug: Dapivirine Gel 4750, 0.05%, 2.5g
- B (Experimental)
  Interventions: Drug: Dapivirine Gel 4789, 0.05%, 2.5g
- C (Placebo Comparator)
  Interventions: Drug: HEC-based Placebo Gel

INTERVENTIONS:
Drug: Dapivirine Gel 4750, 0.05%, 2.5g — intravaginal gel, dosed daily
  Arms: A
Drug: Dapivirine Gel 4789, 0.05%, 2.5g — intravaginal gel, dosed daily
  Arms: B
Drug: HEC-based Placebo Gel — intravaginal gel, dosed daily
  Arms: C

SUMMARY:
IPM 012 is a double-blind, randomized, placebo-controlled phase I study conducted at one research center in Belgium among 36 healthy, HIV-negative women of 18-40 years of age, randomized in a 1:1:1 ratio to assess plasma, vaginal fluid and vaginal tissue levels and the pharmacokinetics of dapivirine when applying either Dapivirine Gel 4750, 0.05%, 2.5g or Dapivirine Gel 4789, 0.05%, 2.5g intravaginally for 11 days (1 day followed by a 3 day washout period and then 10 consecutive days); and to assess the safety of these gels as compared to the intravaginal HEC-based universal placebo gel.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 40 years of age, inclusive
* Willing and able to give written informed consent
* Available for all visits and consent to follow all procedures
* Healthy, based on medical history, vital signs, physical examination, urinalysis, laboratory evaluations for genital infections and laboratory evaluations for hematology, liver and renal function
* HIV-negative as determined by a HIV-1 ELISA test at enrollment
* Willing to abstain from sexual activity for the duration of the study
* On stable oral contraceptive regimen for 2 months prior to enrollment and willing to continue
* Upon pelvic/speculum examination, the cervix and vagina appear normal
* Willing to refrain from the use of vaginal products from 14 days prior to enrollment and for the duration of the study

Exclusion Criteria:

* History of alcoholism, drug abuse, psychosis, antagonistic personality, poor motivation or other emotional or intellectual problems that are likely to invalidate the informed consent process or adversely impact adherence with protocol requirements
* History of sensitivity/allergy to any component of the study product or to latex
* Currently pregnant or breast-feeing, or within 3 months of last pregnancy outcome
* Currently or within one month of participating in any other clinical research study
* History or current diagnosis and/or treatment for a STD within the last three months prior to enrollment
* Current vulvar, vaginal or cervical symptoms/abnormalities as determined by pelvic/speculum exam or colposcopy that could influence the study results
* History of significant urogenital or uterine prolapse, undiagnosed vaginal bleeding or urethral obstruction within the last 3 months
* Current non-iatrogenic pelvic/colposcopic exam findings involving deep epithelial disruption
* Smoking more than 10 cigarettes a day

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Serial dapivirine concentrations in plasma, vaginal fluid and cervical-vaginal tissue samples | 11 days
Self-reported genital symptoms, pelvic/colposcopic exam findings, laboratory evaluations and adverse events/serious adverse events | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Annalene Nel, Study Director — Beijing Immupeutics Medicine Technology Limited
Locations (1):
- SGS Life Science Services Research Unit Stuivenberg, Antwerp, Belgium

REFERENCES:
- [Result] Nel A, Smythe S, Habibi S, Romano J. 2009. Comparison of Safety and PK of Two Formulations of Dapivirine Vaginal Gel in Healthy, HIV-Negative Women [abstract]. 16th Conference on Retroviruses and Opportunistic Infections; 2009 Feb 8-11; Montreal. Available from: http://www.retroconference.org/2009/PDFs/1065.pdf